CLINICAL TRIAL: NCT05179044
Title: Utilization of a Knee Brace With Extension Swing Assist Peri-operatively to Prevent Flexion Contractures and Improves Quadriceps Strength After Total Knee Arthroplasty (TKA)
Brief Title: Utilization of a Knee Brace With Extension Swing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistic difficulties and loss of support from bracing company.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-00143
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Guardian knee brace group (Experimental): Patients undergoing elective Total knee arthroplasty (TKA) by surgeons from NYU Langone with the presence of a pre-operative knee flexion contracture greater than 5 degrees and willingness to participate in our institution's outpatient rehabilitation and physical therapy. Those randomized to this group will be fitted with a Guardian Rehabilitator Brace.
  Interventions: Device: Guardian Sport Rehabilitator knee brace
- No Guardian brace used group (No Intervention): Patients undergoing elective Total knee arthroplasty (TKA) by surgeons from NYU Langone with the presence of a pre-operative knee flexion contracture greater than 5 degrees and willingness to participate in our institution's outpatient rehabilitation and physical therapy as part of standard of care.

INTERVENTIONS:
Device: Guardian Sport Rehabilitator knee brace — The Guardian Sport Rehabilitator knee brace has pneumatic condyles that can be used to support and control the knee joint as well as an extension swing assist design which automatically assists in extending the knee when the patient themselves may guard against it. The Guardian Rehabilitator Knee Brace is considered by the FDA as a Class I external medical device. It is used on label and therefore exempt from IDE requirements.The Guardian Brace FDA registration to manufacturer external limb devices is attached for reference.
  Arms: Guardian knee brace group

SUMMARY:
The purpose of this research is to help determine if use of the Guardian brace during prehab and post-op rehab after TKA can help improve functional outcomes and reduce the incidence of post-operative flexion contractures which reduce knee range of motion after surgery.

DETAILED DESCRIPTION:
This will be a prospective study with consecutive TKA patients with pre-operative flexion contractures of 5 degrees or greater. Patients will be randomized to one of two groups: 1) use of the Guardian knee brace peri-operatively, and 2) no Guardian brace use.

Pre-operative range of motion (ROM) and leg strength will be tested (4 to 6 weeks pre-operatively and the week before surgery) as well as during the recovery period at 6 weeks and 3 months post-operatively. The study will attempt to quantify quadriceps and hamstring strength using a Medical Engineering TKR2000, which can digitally measure quadriceps and hamstring strength with accuracy equivalent to a Biodex Dynanometer. The TKR2000 also accurately measures terminal flexion and extension of the lower extremity. Pre- and post-operative patient reported outcome measures (KOOS JR. score) will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* Surgical candidates undergoing primary TKA
* Surgical candidates with pre-operative flexion contracture of 10 degrees or greater
* Patient is willing to cooperate and follow study protocol and visit schedule

Exclusion Criteria:

* Patient is pregnant
* Patient is unable to provide written consent
* Patient has psychiatric disorder that precludes safe study participation
* Patients with a prior history of surgery in the affected knee
* Vulnerable patient populations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in extensor leg strength | Visit 1( 1 week pre surgery), Visit 2 (2 weeks post surgery) , Visit 3 (6 weeks post surgery), Visit 4 ( 12 weeks post surgery)
  Measured by the TKR2000 which is a patient controlled mechanical over-pressure stretching and strengthening device designed and developed to diminish issues with muscle guarding. The device uses a lever arm with a comfortable foam roller padding placed against the patients' ankle and is moved by an electric actuator. At each scheduled visit, subjects will be examined to determine extensor leg strength on the affected leg.
Change in flexor leg strength | Visit 1( 1 week pre surgery), Visit 2 (2 weeks post surgery) , Visit 3 (6 weeks post surgery), Visit 4 ( 12 weeks post surgery)
  Measured by the TKR2000 which is a patient controlled mechanical over-pressure stretching and strengthening device designed and developed to diminish issues with muscle guarding. The device uses a lever arm with a comfortable foam roller padding placed against the patients' ankle and is moved by an electric actuator. At each scheduled visit, subjects will be examined to determine flexor leg strength on the affected leg.
Change in range of motion following knee replacement surgery | Visit 1( 1 week pre surgery), Visit 2 (2 weeks post surgery) , Visit 3 (6 weeks post surgery), Visit 4 ( 12 weeks post surgery)
  At each scheduled visit, subjects will be examined to determine their range of motion (ROM) in the affected leg to see the range of motion change from pre-op to post- op.

CONTACTS AND LOCATIONS:
Overall Officials: Morteza Meftah, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to daniel.waren@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.